CLINICAL TRIAL: NCT00435656
Title: Pharmacogenetics of Antiretroviral Drugs
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Laure Elens, PhD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: 2006/11OCT/AC/189
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: HIV Infections
Keywords: Human immunodeficiency virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
In this research project, we will study the genetic determinants that influence the pharmacokinetics of antiretroviral drugs used in the treatment of diseases caused by the HIV.

DETAILED DESCRIPTION:
The development of new active substances is a continuous source of progress in pharmacotherapy. However, the search for an optimal use of existing molecules constitutes another possible way of progress. In the particular field of anti-infectious therapy, an optimization of treatments could minimize the emergence of resistance phenomena that require the continuous development of new active molecules.

Pharmacogenetics is the scientific discipline seeking to improve the response to drug therapies (better clinical efficiency and reduction of side effects) by taking into consideration the genetic characteristics of the patient. Drugs with a narrow therapeutic index constitute a main target of this emerging field. The combination of therapeutic drug monitoring and pharmacogenetics already allows to optimize the use of some drugs among which oral anticoagulants, immunosuppressants, antiepileptics, antidepressors, antibiotics or antivirals….

In this research project, we will study the genetic determinants that influence the pharmacokinetics of antiretroviral drugs used in the treatment of diseases caused by the HIV. We will put a particular emphasis on viral protease inhibitors (atazanavir, saquinavir, lopinavir, ritonavir)and non-nucleosides reverse transcriptase inhibitors (nevirapine and efavirenz). For those drugs, the clinician often faces a double therapeutic risk, either of insufficient dosing (clinical inefficacy and emergence of resistance) or of excessive dosing (toxicity). The optimization of drug dosing is especially crucial because some of these drugs often represent the last choice in multi-resistant patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Haufroid, PharmD PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires saint Luc, Brussels, Belgium